CLINICAL TRIAL: NCT05842811
Title: An Observational Study of Patients With Metabolic Syndrome and Related Conditions
Status: Not yet recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-METABOLIC
Record Dates: First submitted 2023-03-09; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood with serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Cohort: Observational
- Engaged Cohort: Observational

SUMMARY:
TARGET-METABOLIC is an observational research study to conduct a comprehensive review of outcomes for patients with metabolic syndrome and related conditions.

ELIGIBILITY:
Disease Cohort

Inclusion Criteria:

- Adult patients at the time of enrollment with a diagnosis of metabolic syndrome or related conditions by ICD-10 code or with clinically calculated BMI ≥ 30 in the EHR/health system interface

Exclusion Criteria:

* Death
* Manual removal (sponsor or site request)
* No EHR interface encounter > 3 years

Engaged Cohort

Inclusion Criteria:

* Adult patients diagnosed and managed for these conditions invited to participate
* Ability to provide written informed consent

Exclusion Criteria:

* Patient expressed desire to withdraw consent to complete PROs
* Failure to complete PROs within 24 weeks of initial invitation
* Greater than 24 months lapse of survey completion after baseline surveys completed
* Additionally, the criteria detailed for Disease Cohort apply to the Engaged Cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults with metabolic syndrome and related conditions.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2023-05-24 (Estimated); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of disease in patients with metabolic syndrome and related conditions | 15 Years
  A detailed analysis of available demographics, anthropometric characteristics, glycemic metrics, medications, co-morbidities, and medical history from sites across the US will inform the profile for various patient populations enrolled into the study. Collection of detailed medical records will be curated and analyzed to characterize disease natural history, clinical course of disease, number and types of interventions, current treatment paradigms, and the patient diagnostic journey. These data may also establish incidence rates of events of special interest. Collection of prospective medical records for each patient enables the continuation of these analyses longitudinally for changes and progression to characterize the clinical course of disease. The progression of pre-existing co-morbidities and variances across populations will also be evaluated.
To assess safety and effectiveness of treatments for metabolic syndrome and related conditions. | 15 Years
  The study will evaluate the characteristics of patients receiving various treatments, effectiveness of treatment, and medical events that develop while receiving treatment for metabolic syndrome and related conditions. Treatments may be pharmacologic, surgical, procedures, radiologic or other interventions given to change the disease course/outcomes. Interval disease and medical events may vary depending on the patient's stage and type of disease and extent of co-morbidities at study entry and time of diagnosis.

SECONDARY OUTCOMES:
To evaluate provider management practices in the treatment of patients with metabolic syndrome and related conditions | 15 Years
  Health care provider type, clinic setting, reason for initiating/not initiating/adjusting dosing of treatments or interventions (i.e., surgery, radiation), reason for discontinuing/switching treatments, and monitoring outcomes on and off treatment, will be captured as available in the provided EHR and/or through linked data. Disease-specific quality measures will be selected and evaluated, and the curated data can enable analyses to describe and evaluate healthcare utilization patterns.
To evaluate longitudinal and patient reported outcomes in patients with metabolic syndrome and related conditions | 15 Years
  Longitudinal clinical outcomes and disease progression will be assessed. Self-reported patient health measures collect information directly from patients to measure physical, mental, and social health. These measures can help clinicians better understand how the disease state and/or various treatments affect what patients are able to do and the symptoms they experience beyond what is typically derived and reported in the EHR as part of traditional clinical evaluations. The information can also be used to help patients make informed decisions about their healthcare and treatment options.
To select and evaluate quality of care measures for patients with metabolic syndrome and related conditions | 15 Years
  1. Identify deficiencies and select best practices in care of patients
  2. Develop a technology infrastructure to evaluate quality measures to support clinicians.

IPD SHARING:
Plan to Share IPD: Undecided